CLINICAL TRIAL: NCT04185467
Title: The Effectiveness of Rehabilitation for Patients With Lung Cancer in China: a Randomised Controlled Trial
Brief Title: Lung Cancer Rehabilitation After Medical Treatment
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The coronavirus broke out in China at the end of 2019
Sponsor: Nantong University (Other)
Collaborators: University of Melbourne (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jun Ni, Director of Rehabilitation Treatment Center, Nantong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NantongU
Record Dates: First submitted 2019-11-23; First posted 2019-12-04 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Lung Neoplasms
Keywords: lung cancer; exercise; rehabilitation; Tai Chi; health-related quality of life
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Methods; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Design: Two-site, assessor blinded, two-arm superiority randomised controlled trial.
  Setting: Participant recruitment from the affiliated hospital of Nantong University and the first affiliated hospital of Nanjing Medical University
  Procedure:
  Randomisation: Randomisation list devised by independent statistician; carried out using the REDCap randomisation function to ensure allocation concealment. Following consent and assessment, participants are randomised 1:1. Lung cancer with stage I-IIIA and treatment type is surgery +/- adjuvant treatment.
Who Masked: Outcomes Assessor
Masking Description: Assessor blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care(both arms) (No Intervention): Usual care (both arms): Patients in both arms will receive usual medical, physiotherapy and nursing care according to usual protocols. This does not involve exercise rehabilitation or advice.
- Intervention (exercise rehabilitation) (Experimental): Patients in intervention group (exercise rehabilitation) will receive a multimodal program which includes a 90 minute program at the hospital gymnasium in a supervised environment a minimum of once but up to twice per week. Rehabilitation will include aerobic (brisk walking), resistance training and 30 minutes of 8 style Tai Chi. Participants will be advised to walk on days of non-attendance - this will be individualised with the aim to have participants increase to 30 minutes walking per day.
  Interventions: Other: Intervention (rehabilitation exercise)

INTERVENTIONS:
Other: Intervention (rehabilitation exercise) — Patients in intervention group (exercise rehabilitation) will receive a multimodal program which includes a 90 minute program at the hospital gymnasium in a supervised environment a minimum of once but up to twice per week. Rehabilitation will include aerobic (brisk walking), resistance training and 30 minutes of 8 style Tai Chi. Participants will be advised to walk on days of non-attendance - this will be individualised with the aim to have participants increase to 30 minutes walking per day.
  Arms: Intervention (exercise rehabilitation)

SUMMARY:
Lung cancer is the leading cause of cancer death worldwide and associated with high disease burden, symptoms and poor health-related quality of life (HRQoL). Lung cancer is the most commonly diagnosed type of cancer in China (with rates rising due to the smoking incidence) and is the leading cause of cancer-related death. The burden is on patients, families, the healthcare system and society, and will continue to rise into the future. The full impact of this in China has not yet occurred. New strategies are urgently required to improve survivorship. This multi-site, assessor blinded, two-arm superiority randomised controlled trial, conducted at two hospitals in China, aims to test the effect of exercise rehabilitation, compared to usual care (no exercise rehabilitation) on HRQoL and functional outcomes in 150 patients treated for lung cancer. The primary hypothesis is that exercise rehabilitation will be superior to usual care, in improving HRQoL at 12-weeks (post program). Secondary aims include measuring the effectiveness of exercise rehabilitation, compared to usual care on function, physical activity, symptoms, mood, sleep and program costs. Faecal samples (500mg) will be collected before and after the intervention.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death worldwide and associated with high disease burden, symptoms and poor health-related quality of life (HRQoL). Lung cancer is the most commonly diagnosed type of cancer in China (with rates rising due to the smoking incidence) and is the leading cause of cancer-related death. The burden is on patients, families, the healthcare system and society, and will continue to rise into the future. The full impact of this in China has not yet occurred. New strategies are urgently required to improve survivorship. This multi-site, assessor blinded, two-arm superiority randomized controlled trial, conducted at two hospitals in China, aims to test the effect of exercise rehabilitation, compared to usual care (no exercise rehabilitation) on HRQoL and outcomes including physical function in 150 patients treated for lung cancer. The primary hypothesis is that exercise rehabilitation will be superior to usual care, in improving HRQoL at 12-weeks (post program). Secondary aims include include measuring the effectiveness of exercise rehabilitation, compared to usual care on function, physical activity, symptoms, mood, sleep and program costs.

One hundred and fifty patients with stage I-IIIA non-small cell lung cancer (NSCLC) 4-12 weeks following completion of treatment (including surgery with or without adjuvant therapy) and life expectancy greater than 6 months will be recruited from the affiliated hospital of Nantong University and the first affiliated hospital of Nanjing Medical University. At recruitment participants provide written informed consent, complete baseline assessment and to ensure concealment of allocation participants will be randomly allocated off-site to one of two arms (1:1 ratio). The intervention programs start following randomization and will continue for 12 weeks duration. Trained physiotherapists will provide the intervention. Patients in both arms will receive usual medical, physiotherapy and nursing care according to usual protocols. This does not involve exercise rehabilitation or advice. Additionally patients in intervention group (exercise rehabilitation) will receive a multimodal program which includes a 90 minute program at the hospital gymnasium in a supervised environment a minimum of once but up to twice per week. Rehabilitation will include aerobic (brisk walking) and resistance training and 30 minutes of 8 style Tai Chi). Participants will be advised to walk on days of non-attendance - this will be individualized with the aim to have participants increase to 30 minutes walking per day. Assessments will be conducted at baseline and then by blinded assessors at 12 weeks and 6 months post-baseline. Survival will be followed-up and censored at 1 year. This important study brings together a strong collaborative research team spanning China and Australia, involving medical doctors, physiotherapists and academics. The topic is important, novel and will generate clinically meaningful research for an international audience, aiming to improve the survivorship quality of patients with lung cancer.

The gut microbiome is a source of potentially disease-modifying bioactive metabolites and has recently been suggested to contribute to the pathogenesis of a variety of disorders. Therefore, we will study the gut microbiota and metabolites of the participants in order to identify potential the biomarkers for the clinical outcomes. Fresh faecal samples will be collected from all individuals before group assignment and after the completion of the program. The written informed consent will be provided by the participants.

Specifically, faecal samples (500mg) will be collected from participants who are free from gastrointestinal conditions, with no antibiotic exposure in the 28 days prior to sample collection. 'Snap' frozen samples will be stored at -80°C until the time of DNA extractions, 16S rDNA sequencing, and mass spectrometry analysis of the faecal metabolites. The distribution of gut microbiota before and after exercise will be compared and analyzed to obtain the species of bacterial flora that changed significantly after exercise. Moreover, the gut metabolites that changed significantly before and after exercise will be used to explore the biomarkers for the curative effect of rehabilitation exercise, as well as their relationships with the differentially distributed gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-small cell lung cancer (NSCLC) 4-12 weeks following completion of treatment (surgery, chemotherapy, radiotherapy, immunotherapy);
2. Physician/doctor approval;
3. Physician rated life expectancy greater than 6 months;
4. Informed consent;
5. Eastern Cooperate Oncology Group (ECOG) performance status of 0-2 at study entry;
6. Not meeting physical activity/exercise guidelines.

Exclusion Criteria:

1. Unstable psychiatric/cognitive disorder;
2. Comorbidity preventing exercise;
3. ECOG performance status of 3 or 4 at study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
European Organization for the Research and Treatment of Cancer questionnaire (EORTC QLQ-C30-LC13) | The primary time point is the change from baseline to 12 weeks. This outcome will also be measured at 6 months post-baseline.
  HRQoL will be assessed with the European Organization for the Research and Treatment of Cancer questionnaire (EORTC QLQ-C30-LC13) at baseline, 12 weeks and 6 months post-baseline. Score ranges from 0~100.For functional domains and global health status/quality of life scale, higher score means better status. While for symptom domains and single-items, lower scores represent less symptoms.

SECONDARY OUTCOMES:
Functional Exercise Capacity | 1) baseline, 2) 12 week, and 3) 6 months post-baseline.
  All participants will complete a Incremental Shuttle Walking Test following published guidelines.
Seven-day Physical Activity | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  Will be measured objectively using an pedometer at baseline, 12 weeks and 6 months post-baseline. It is worn for 7 consecutive days and a minimum of four full days (8 hours/day) is required for valid analyses.
Grip strength | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  A hand held dynamometry manual muscle test is a common, simple measurement of strength and has been used in many patient populations including cancer and is reliable and sensitive to change. We will measure hand grip strength bilaterally
30-Second Chair Stand | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  To test leg strength and endurance. A below average score indicates a risk for falls.
International physical activity questionnaire(IPAQ) | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  The International Physical Activity Questionnaire (IPAQ) scores are categorised as high/moderate (meeting PA guidelines) or low (not meeting PA guidelines) and as a continuous energy expenditure score (metabolic equivalent of task (MET) minutes per week). Higher scores indicate increased PA.
Self-Rating Anxiety Scale(SAS) | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  To test the anxiety level of the patients. It has 20 items and are four-point scale(rated 1-4), some of the items are reversely scored. Score ranges from 0~100, higher score means worse anxiety status.
Self-Rating Depression Scale(SDS) | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  To test the depression level of the patients. It has 20 items and are four-point scale(rated 1-4), some of the items are reversely scored. Score ranges from 0~100, higher score means worse depression status.
Pittsburgh Sleep Quality Index(PSQI) | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  Pittsburgh Sleep Quality Index(PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores. The sum of scores for these seven components yields one global score, and the higher score means the worse sleep quality. Score ranges from 0~21, higher score means worse sleep quality.
MD Anderson Symptom Inventory-lung cancer (MDASI-LC) | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  To evaluate to the severity and interference of the symptom in participants.The MD Anderson Symptom Inventory-Lung Cancer (MDASI-LC) will be used to measure symptom severity and distress. The symptom severity component comprises 13 core and three lung cancer specific items, measured on a 0-10 numerical rating scale. The average score is reported, with higher scores indicating worse symptoms. The MCID in lung cancer has been reported as being between 0.98 to 1.21 points
Australia-modified Karnofsky Performance Status(AKPS) | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  To evaluate the performance of the whole well-being of the participants. Score ranges from 0~100, higher score means better status.
European quality of life 5-dimension 5-level(EQ-5D-5L) | 1) baseline, 2) 12 weeks, and 3) 6 months post-baseline.
  European quality of life 5-dimension 5-level(EQ-5D-5L) is a family of instruments to describe and value health. It comprises a short descriptive system questionnaire and a visual analogue scale that are cognitively undemanding. A value set provides values(weights) for each health state description according to the preferences of the general population of a country/region.

OTHER OUTCOMES:
Adherence to the program | 12 weeks post-program
  Intervention group participants who complete either 17 out of 24 hospital-sessions or 12 out of 24 hospital sessions and at least 10 minutes walking at home twice a week will be considered to be adherent to the protocol.
Program costs | Baseline, 12 weeks (post-program) and 6 months
  We will consider the additional implementation costs of rehabilitation, including patient costs, compared with usual care in addition to the downstream cost differences associated with hospital usage (including hospital admissions and their length of stay, visits to accident and emergency and clinic appointments). Health from baseline to 6 months (with modelling to 12 months) will be measured using Quality Adjusted Life Years (QALYs) and then within trial follow-up cost per additional QALY will be estimated and compared with levels considered to provide good value for money. Probabilistic sensitivity analysis will be conducted to explore the robustness of the conclusions reached.
Survival | 12 months post baseline
  We will follow up survival in all groups and censor at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ni, MD, Principal Investigator — Nantong University
Locations (2):
- China (2):
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - the Affiliated Hospital of Nantong University, Nantong, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available to other investigators for individual participant data meta-analysis.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Hung R, Krebs P, Coups EJ, Feinstein MB, Park BJ, Burkhalter J, Ostroff JS. Fatigue and functional impairment in early-stage non-small cell lung cancer survivors. J Pain Symptom Manage. 2011 Feb;41(2):426-35. doi: 10.1016/j.jpainsymman.2010.05.017. Epub 2011 Jan 8. PMID 21216563
- [Background] Hong QY, Wu GM, Qian GS, Hu CP, Zhou JY, Chen LA, Li WM, Li SY, Wang K, Wang Q, Zhang XJ, Li J, Gong X, Bai CX; Lung Cancer Group of Chinese Thoracic Society; Chinese Alliance Against Lung Cancer. Prevention and management of lung cancer in China. Cancer. 2015 Sep 1;121 Suppl 17:3080-8. doi: 10.1002/cncr.29584. PMID 26331814
- [Background] Polanski J, Jankowska-Polanska B, Rosinczuk J, Chabowski M, Szymanska-Chabowska A. Quality of life of patients with lung cancer. Onco Targets Ther. 2016 Feb 29;9:1023-8. doi: 10.2147/OTT.S100685. eCollection 2016. PMID 27013895
- [Background] Zhang LL, Wang SZ, Chen HL, Yuan AZ. Tai Chi Exercise for Cancer-Related Fatigue in Patients With Lung Cancer Undergoing Chemotherapy: A Randomized Controlled Trial. J Pain Symptom Manage. 2016 Mar;51(3):504-11. doi: 10.1016/j.jpainsymman.2015.11.020. Epub 2015 Dec 22. PMID 26721747
- [Background] John LD. Self-care strategies used by patients with lung cancer to promote quality of life. Oncol Nurs Forum. 2010 May;37(3):339-47. doi: 10.1188/10.ONF.339-347. PMID 20439218
- [Background] Schmitz KH, Holtzman J, Courneya KS, Masse LC, Duval S, Kane R. Controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. Cancer Epidemiol Biomarkers Prev. 2005 Jul;14(7):1588-95. doi: 10.1158/1055-9965.EPI-04-0703. PMID 16030088
- [Background] Lin YY, Rau KM, Lin CC. Longitudinal study on the impact of physical activity on the symptoms of lung cancer survivors. Support Care Cancer. 2015 Dec;23(12):3545-53. doi: 10.1007/s00520-015-2724-7. Epub 2015 Apr 9. PMID 25855040
- [Background] Wang JW, Gong XH, Ding N, Chen XF, Sun L, Tang Z, Yu DH, Yuan ZP, Wang XD, Yu JM. The influence of comorbid chronic diseases and physical activity on quality of life in lung cancer survivors. Support Care Cancer. 2015 May;23(5):1383-9. doi: 10.1007/s00520-014-2494-7. Epub 2014 Oct 31. PMID 25358644
- [Background] Jones LW, Watson D, Herndon JE 2nd, Eves ND, Haithcock BE, Loewen G, Kohman L. Peak oxygen consumption and long-term all-cause mortality in nonsmall cell lung cancer. Cancer. 2010 Oct 15;116(20):4825-32. doi: 10.1002/cncr.25396. PMID 20597134
- [Background] Brown JC, Schmitz KH. The prescription or proscription of exercise in colorectal cancer care. Med Sci Sports Exerc. 2014 Dec;46(12):2202-9. doi: 10.1249/MSS.0000000000000355. PMID 24781887
- [Background] Gopalakrishnan V, Helmink BA, Spencer CN, Reuben A, Wargo JA. The Influence of the Gut Microbiome on Cancer, Immunity, and Cancer Immunotherapy. Cancer Cell. 2018 Apr 9;33(4):570-580. doi: 10.1016/j.ccell.2018.03.015. PMID 29634945
- [Background] Keohane DM, Woods T, O'Connor P, Underwood S, Cronin O, Whiston R, O'Sullivan O, Cotter P, Shanahan F, Molloy MGM. Four men in a boat: Ultra-endurance exercise alters the gut microbiome. J Sci Med Sport. 2019 Sep;22(9):1059-1064. doi: 10.1016/j.jsams.2019.04.004. Epub 2019 Apr 18. PMID 31053425
- [Background] Hamasaki H. Exercise and gut microbiota: clinical implications for the feasibility of Tai Chi. J Integr Med. 2017 Jul;15(4):270-281. doi: 10.1016/S2095-4964(17)60342-X. PMID 28659231